CLINICAL TRIAL: NCT01399463
Title: Pressure Wire-guided Percutaneous Coronary Intervention of Small Vessels or Side Branches: Functional Outcome of Drug-Eluting Stent (DES) Versus Drug-Eluting Balloon (DEB) With Provisional Bare Metal Stent Implantation
Brief Title: Pressure-wire Guided PTCA: Drug Eluting Stent Versus Drug Eluting Balloon (WinDEB Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Thomas Neunteufl, MD, Univ. Klinik für Innere Medizin II; Department of Cardiology
Model: Parallel | Masking: Single
Other Study IDs: MUWCard18022011
Record Dates: First submitted 2011-07-20; First posted 2011-07-21 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Coronary Artery Disease
Keywords: Drug Eluting Stent, Drug Eluting Balloon, Fractional Flow Reserve, DES, DEB, FFR
MeSH Terms: conditions — Coronary Artery Disease; Dysequilibrium syndrome

ARMS (2):
- DEB + BMS (Experimental): Paclitaxel drug-eluting balloon (DEB) dilatation and bare metal stenting
  Interventions: Device: Angioplasty performed via Paclitaxel Eluting Balloon catheter
- Stenting with commonly used Drug Eluting Stents (DES) (Active Comparator)
  Interventions: Device: Angioplasty via DES

INTERVENTIONS:
Device: Angioplasty performed via Paclitaxel Eluting Balloon catheter
  Arms: DEB + BMS
Device: Angioplasty via DES — Angioplasty performed via commonly used Drug Eluting Stents
  Arms: Stenting with commonly used Drug Eluting Stents (DES)

SUMMARY:
The aim of the study is to show the safety and efficacy of the SeQuent® Please (Drug Eluting Balloon or DEB) vs. commonly used Drug Eluting Stents in the treatment of small vessel disease and side branches by pressure wire guided percutaneous coronary intervention.

DETAILED DESCRIPTION:
This study is a randomized, prospective, multi-center, efficacy study with a DES control group assessing the 6-month loss in FFR in patients treated with the "matrix coated paclitaxel-eluting PTCA-balloon catheter" SeQuent® Please and commonly used DES for small vessel de novo and side branch lesions. 100 patients will be studied in total with two equivalent treatment groups DEB & DES of 50 patients each.

ELIGIBILITY:
Inclusion Criteria:

* Patients of at least 18 years of age.
* Patients with stable angina pectoris (CCS class 1-3) or with unstable angina pectoris (Braunwald class 1-2, A-C) or documented ischemia or with documented silent ischemia
* Patients must agree to undergo the angiographic 6-month and clinical follow-ups at 12 and 36 months.
* De novo coronary lesions including side branches in native coronary arteries (reference vessel between ≥ 2.0 and ≤ 3.0 mm, lesion length ≤ 25 mm as angiographically documented)
* Diameter stenosis pre procedure must be either ≥ 70 % or ≥ 50 % if ischemia corresponding to the target lesion is documented either by exercise stress ECG, stress echocardiography, scintigraphy, MRT, or suspected based on angina pectoris.
* Fractional Flow Reserve (FFR) must be less or equal to 0.75.

Exclusion Criteria:

* Patients with a life expectancy of less than 12 months
* Patients that were treated with one or more DES during the last 12 months which would not allow 3-month dual antiplatelet therapy if the patient were randomized in the DEB treatment group.
* Patients who are obliged to be on dual antiplatelet aggregation therapy for more than 3 months following study inclusion
* Patients with acute (< 24 h) or recent (48 hours) myocardial infarction
* Patients with severe congestive heart failure or with severe heart failure NYHA IV or with severe valvular heart disease
* Patients demonstrating clinical signs of cardiogenic shock at the time of the procedure (systolic blood pressure of less than 80 mmHg requiring inotropic support, IABP and/or fluid challenge)
* DES treated lesion(s) during the last 12 months.
* Thrombus burden (STEMI, NSTEMI) and/or total occlusion in the culprit segment
* In-segment stenosis of the native vessel within the 5 mm adjacent to the stent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2011-08

PRIMARY OUTCOMES:
Loss in fractional flow reserve (FFR) at 6 months for both treatment groups | 6 month

SECONDARY OUTCOMES:
Occurrence of acute (up to 48 hours), subacute (up to 30 days) and late stent thrombosis | acute: <48h; subacute: < 30days
NACCE rate at 30 days, 6 and 12 months | 30days, 6 and 12 month
Procedural success
Percent in-stent stenosis, in-segment stenosis, in-stent late lumen loss and in-segment late lumen loss at 6 months follow-up | 6 month
  Percent in-stent stenosis, in-segment stenosis, in-stent late lumen loss and in-segment late lumen loss at 6 months follow-up
Angiographic in-stent restenosis rate of the target lesion (≥ 50 % stenosis) at 6 months from the procedure | 6 month
Angiographic in-segment stenosis rate of the target lesion (≥ 50 % stenosis) at 6 months from the procedure | 6 month
Indication for premature follow-up
Target vessel failure